CLINICAL TRIAL: NCT06098534
Title: Evaluation d'un Prototype de Chambre Innovante adaptée au Grand Age
Brief Title: Evaluation of a Prototype for an Innovative Room for the Elderly
Acronym: HOSPISENIOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 49RC23_0276
Record Dates: First submitted 2023-10-11; First posted 2023-10-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Elderly Inpatients
Keywords: Prototype; Care; Hospital Room; Elderly; Innovation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Hospi'Senior" group (Experimental): Patients admitted to the Hospi'Senior room benefit from the innovative technologies available in this room. Patients benefit from standard care throughout their hospital stay.
  Interventions: Behavioral: Hospi'Senior
- "Conventional room" group (Experimental): Patients admitted to a conventional room receive the standard care throughout their hospital stay.
  Interventions: Behavioral: Conventional room

INTERVENTIONS:
Behavioral: Hospi'Senior — The Hospi'Senior room is equipped with conventional furnishings (same bed and same armchair as a conventional room) to which have been added technological innovations and innovations in furnishings. Innovative technologies cover bed equipment, patient mobility (autonomous and assisted), lighting, communication and social space.
  Arms: "Hospi'Senior" group
Behavioral: Conventional room — The conventional room is a classic hospital room not equipped with the innovative technologies found in the Hospi'Senior room.
  The room is equipped with a bed, bedside table, adjustable bed table with castors and an armchair.
  Arms: "Conventional room" group

SUMMARY:
The Groupement de Coopération Sanitaire des Hôpitaux Universitaires du Grand Ouest (GCS HUGO) (health cooperation group for university hospitals in the west of France), is proposing to improve the quality of geriatric care by modernizing hospital rooms. The GCS HUGO has embarked on a project to co-design a hospital room adapted for the elderly, called "Hospi'Senior", with the help of the "Dépendance et Grand âge" (Dependency and Old Age) steering committee, made up of experts from HUGO's establishments and experts from several companies.

DETAILED DESCRIPTION:
The main objective is to evaluate the effect of hospitalization in a Hospi'Senior room on the length of stay of elderly people compared with hospitalization in a conventional room for a similar admission reason.

The secondary objectives are to evaluate the effect of hospitalization in a Hospi'Senior room for elderly people, compared with hospitalization in a conventional room for a similar admission reason, on :

2) Changes in functional abilities during the hospital stay and in the 30 days following discharge from the short-stay geriatric unit 3) Occurrence of behavioral disorders 4) Occurrence of falls during the hospital stay and in the 30 days following discharge from the short-stay geriatric unit 5) Occurrence and/or worsening of stage bedsores ≥ 2 during the hospital stay as classified by the National Pressure Ulcer Advisory Panel (NPUAP) 6) Occurrence of early rehospitalization

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Admission in a short-stay geriatric department following initial emergency care department or direct entry from home
* Hospitalization in single room: Hospi'Senior or conventional
* Affiliation to a social security scheme
* Informed consent to participate in the study from the patient or his/her representative (tutor/curator if applicable, or in order of priority a trusted person, the family or a person with whom the person concerned has a close and stable relationship)

Exclusion Criteria:

* Contraindication to study participation at the discretion of the medical team
* Hospitalization for more than 3 days (>3 days) in the short-stay geriatric unit
* Hospitalization in a double room
* Planned hospitalization
* Poor understanding of the French language
* Patient under safeguard of justice

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-11-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Length of stay in the short-stay geriatric unit | This outcome is assessed at the end of the geriatric unit stay (up to 2 months)
  The length of stay is measured in days

SECONDARY OUTCOMES:
Changes in functional capabilities | This outcome is assessed at inclusion, on discharge (up to 2 months) and within 30 days of discharge from the short-stay geriatric unit
  Functional capabilities are assessed with Activities of Daily Living (ADL) score.
  ADL is an autonomy assessment grid (from 0 to 6) for basic activities of daily living. The lower the score, the more dependent the patient is.
Occurrence of behavioral disorders | This outcome is assessed at inclusion and on discharge (up to 2 months)
  Behavioral disorders are assessed with Neuropsychiatric Inventory-nursing home version (NPI-NH) score.
  For each scale domain, higher scores indicate greater neuropsychiatric symptomatology (range from 0 to 12/12).
Occurrence of falls | This outcome is assessed on discharge (up to 2 months) and within 30 days of discharge from the short-stay geriatric unit
  Number of falls observed during hospital stay and within 30 days of discharge from the short-stay geriatric unit
Occurrence and/or worsening of stage bedsores ≥ 2 | This outcome is assessed on discharge (up to 2 months)
  Occurrence and/or worsening of stage bedsores ≥ 2 during hospital stay
Occurrence of early rehospitalization | This outcome is assessed within 30 days of discharge from the short-stay geriatric unit
  Number of unscheduled hospitalization in a Medicine-Surgery-Obstetrics (MSO) unit within 30 days of discharge from the short-stay geriatric unit

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carcreff L, Briere O, Chapelet G, Fougere B, Gentric A, Somme D, Paolantoni F, Gaudin F, Annweiler C, Noublanche F. User experience of innovative hospital rooms for older patients: the HospiSenior project. Geriatr Psychol Neuropsychiatr Vieil. 2025 Dec 1;23(4):458-467. doi: 10.1684/pnv.2025.1254. PMID 41627010